CLINICAL TRIAL: NCT04948424
Title: A Retrospective Observational Study to Describe Anaemia Management, Burden of Disease and Outcomes in Chinese Patients on Peritoneal Dialysis Using a Clinical Database
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); Army Medical University, China (Other); The First Affiliated Hospital of Zhengzhou University (Other); Hebei Medical University Third Hospital (Other); Peking University Shenzhen Hospital (Other); Handan Central Hospital, Hebei (Unknown); Peking Haidian Hospital (Unknown); People's Hospital of Qinghai Province (Unknown); Cangzhou Central Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Shengjing Hospital (Other); The Second Hospital of Anhui Medical University (Other); Peking University People's Hospital (Other); The First Affiliated Hospital of BaoTou Medical College (Other); The People's Hospital of Chuxiong Yi Autonomous Prefecture (Unknown); Beijing miyun district hospital (Unknown); Second Hospital of Shanxi Medical University (Other); People's Hospital of Gansu (Unknown); Pingdingshan first people's Hospital (Unknown); The first people's hospital of Xining (Unknown); The First Hospital of Jilin University (Other); Cangzhou People's Hospital (Other); Taiyuan central hospital (Unknown); People's hospital of Langfang (Unknown); China Rehabilitation Research Center (Other Government); Dongzhimen Hospital, Beijing (Other); Department of Epidemiology and Biostatistics, School of Public Health, Peking University (Unknown)
Responsible Party: Principal Investigator, Dong Jie, Clinical Professor in Renal Division，Department of Medicine, Peking University First Hospital
Other Study IDs: Anaemia, retrospective
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall objective is to describe the epidemiology, health care resource utilisation (HCRU) and selected clinical outcomes in patients initiating PD by anaemia status in real-world setting in China.

DETAILED DESCRIPTION:
Real-world evidence for chronic kidney disease (CKD)-associated anemia in China is scarce. This study aims to provide supporting novel evidence for the real-world management and treatment of patients on PD with CKD-associated anemia. This is an observational cohort study using secondary data. The data source is the PD Telemedicine-based Management Platform (PDTAP) database, which is a clinical database that prospectively collects data in patients receiving PD and evaluates PD management and clinical practice in China. The PDTAP database has enrolled around 7,000 patients receiving PD from 27 hospitals in 14 provinces located in all seven geographical regions (northwest, northeast, north, central, southwest, southeast and south) in China.

The overall objective is to describe the epidemiology, patient characteristics, treatment patterns relevant to anemia and clinical outcomes in patients on PD in real-world practice in China. Specifically, the incidence and prevalence of anemia will be estimated. The patient characteristics, medication use, select laboratory values and clinical outcomes, and healthcare resource utilization (HCRU) will be described in PD patients with and without anemia. The primary outcomes are 1) the incidence and prevalence of anemia, including the factors that predict the incidence of anemia; 2) the number and percentage of patients who experienced all-cause hospitalizations; 3) adverse clinical outcomes, such as mortality MACE and modified MACE+. The secondary outcomes are 1) hemoglobin levels or anemia, iron variables, medications on anemia management and clinical outcomes in patients with or without inflammation; 2) ESA responsiveness; 3) Other clinical outcomes, such as transfer to hemodialysis and peritonitis.

Associations between anemia, anemia-relevant factors and above clinical outcomes can be analyzed in series of paper with specific aims. For example, 1) the relationship between hemoglobin levels or anemia and clinical outcomes (such as mortality, MACE, modified MACE+, hospitalization, transfer to hemodialysis and peritonitis); 2) prognostic factors that predict the incidence of anemia during the follow up; 3) hemoglobin levels or anemia, iron variables, medications on anemia management and clinical outcomes in patients with or without inflammation; 4) the relationship between hemoglobin levels or anemia, erythropoietin responsiveness and clinical outcomes; 5) prognostic factors that predict the hyporesponsiveness to erythropoietin; 6) determine cut-off values of the iron index (such as serum iron, ferritin, TIBC and TSAT) to predicting worse clinical outcomes. Each study could select hemoglobin relevant variables including clinical characteristics and treatment patterns at baseline and/or during the follow up, and explore their associations with specific clinical outcomes.

Confounding, interaction or mediation effects could be evaluated. Subgroups, such as with or without diabetes, with or without CVD, with or without inflammation status et al could be analyzed as needed. Cox, competing risk models, Poisson or NegBin regression models may be used as needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years old at the initiation of peritoneal dialysis
* Patients with CKD with the first treatment/initiation of peritoneal dialysis between 1 June 2016 and 30 April 2019 with up to 2 years of follow-up data.
* Receiving PD for>3 months

Exclusion Criteria:

* Patients with missing age or sex information (proportion of missingness to be assessed)
* Patients with diagnosises of any cancer (except for non-melanoma skin cancer) within 12 months prior to and inclusive of the baseline date
* Patients with evidence of active bleeding within 30 days and inclusive of the baseline date
* Patients with peritoneal dialysis switched from hemodialysis or renal transplantation failure
* Individuals receiving temporary PD (duration < 30 days) because of acute kidney injury.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is primarily descriptive and all patients meeting the inclusion criteria will be included. We expect to analysis data on approximately 2000 to 2500 peritoneal dialysis patients.
Sampling Method: Probability Sample
Enrollment: 2519 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Anemia | June 1, 2016 to December 31, 2020
  the incidence and prevalence of anemia; factors that predict the incidence of anemia
Healthcare resource utilisation | June 1, 2016 to December 31, 2020
  the number and percentage of patients who experienced all-cause hospitalisations.
Select adverse clinical outcomes | June 1, 2016 to December 31, 2020
  Such as mortality, MACE, modified MACE+

SECONDARY OUTCOMES:
Compare the anemia-related index between patients with and without inflammation | June 1, 2016 to December 31, 2020
  Anemia-related index for participants with and without inflammation
ESA responsiveness | June 1, 2016 to December 31, 2020
  Such as describing trajectories of Hb level and ESA dose post-ESA initiation and explore the relationship among erythropoietin responsiveness, hemoglobin levels and clinical outcomes
Select adverse clinical outcomes | June 1, 2016 to December 31, 2020
  Such as transfer to hemodialysis and peritonitis

CONTACTS AND LOCATIONS:
Overall Officials: Jie Dong, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China